CLINICAL TRIAL: NCT03059420
Title: Genetic Studies of Strabismus, Congenital Cranial Dysinnervation Disorders (CCDDs), and Their Associated Anomalies
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Howard Hughes Medical Institute (Other)
Responsible Party: Principal Investigator, Elizabeth Engle, Investigator, Howard Hughes Medical Institute; Professor of Neurology and Ophthalmology, Harvard Medical School, Boston Children's Hospital
Other Study IDs: 05-03-036R
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Congenital Fibrosis of Extraocular Muscles; Duane Retraction Syndrome; Duane Radial Ray Syndrome; Mobius Syndrome; Brown Syndrome; Marcus Gunn Syndrome; Strabismus Congenital; Horizontal Gaze Palsy; Horizontal Gaze Palsy With Progressive Scoliosis; Facial Palsy; Facial Paresis, Hereditary, Congenital; Third Nerve Palsy; Fourth Nerve Palsy; Sixth Nerve Palsy; Synkinesis; Ocular Motility Disorders; Levator-Medial Rectus Synkinesis; Athabaskan Brainstem Dysgenesis; Tongue Paralysis; Ninth Nerve Disorder; Fifth Nerve Palsy; Seventh Nerve Palsy; Eleventh Nerve Disorder; Twelfth Nerve Disorder; Vagus Nerve Paralysis; Moebius Sequence
Keywords: CFEOM (Congenital Fibrosis of Extraocular Muscles); CCDD (Congenital Cranial Dysinnervation Disorders); DRS (Duane Retraction Syndrome); DRRS (Duane Radial Ray Syndrome); Strabismus; MGJWS (Marcus Gunn Jaw Winking Syndrome); HGP (Horizontal Gaze Palsy); HGPPS (Horizontal Gaze Palsy with Progressive Scoliosis); Moebius
MeSH Terms: conditions — Congenital Cranial Dysinnervation Disorders; Duane Retraction Syndrome; Mobius Syndrome; Ocular Motility Disorders; Marcus Gunn phenomenon; gaze palsy, familial horizontal, with progressive scoliosis; Facial Paralysis; Facial paresis, hereditary, congenital; Oculomotor Nerve Diseases; Trochlear Nerve Diseases; Abducens Nerve Diseases; Synkinesis; Levator-Medial Rectus Synkinesis; Athabaskan brainstem dysgenesis; Glossopharyngeal Nerve Diseases; Bell Palsy; Accessory Nerve Diseases; Hypoglossal Nerve Diseases; congenital fibrosis of the extraocular muscles; Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Following specimens may be submitted: saliva, blood, discarded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify genes associated with impaired development and function of the cranial nerves and brainstem, which may result in misalignment of the eyes (strabismus) and related conditions.

DETAILED DESCRIPTION:
If left untreated or unrecognized, strabismus or misalignment of the eyes, can impair the development of normal vision and is recognized to be an inherited trait in some families. The Engle Lab has investigated the genetics of complex and common strabismus and eyelid movement disorders for over 10 years and the lab's interests have expanded to include Congenital Cranial Dysinnervation Disorders (CCDDs) which are neurological disorders affecting one or more of the 12 cranial nerves. Cranial nerves control bodily functions such as movement of the eyes, transmission of visual information, smell, facial sensation, facial expression, blinking, hearing, balance, taste, chewing and swallowing.

Based on genetic studies on individuals with eye movement and eyelid disorders, the lab learned that some individuals have additional ocular defects, vascular, limb and other abnormalities. In addition, in some families relatives who carry the gene mutation may manifest the familial syndrome by having only some additional features but NOT the oculomotility disorder. Therefore, to gain greater understanding of the spectrum of the disorders being investigated, we may also enroll individuals without eye movement or lid defects who have symptoms associated with mutations in congenital cranial dysinnervation disorder (CCDD) genes.

ELIGIBILITY:
Inclusion Criteria:

* The Engle Lab is very interested in enrolling individuals with congenital conditions related to eye movement, cranial nerve and brainstem-based dysfunction, often broadly referred to as congenital cranial dysinnervation disorders (CCDDs).

Exclusion Criteria:

* Individuals with cranial nerve disorders associated with known disorders, such as Saethre-Chotzen associated with established genetic mutations, or acquired conditions including trauma, stroke, tumor or spinal cord injuries.

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with strabismus, congenital ocular motility disorders, cranial nerve dysfunction, brainstem disorders and other associated anomalies, as well as their similarly affected or unaffected family members. Unaffected individuals are enrolled only if a relative is diagnosed with one of these conditions at least one affected family members is enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2004-02-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Identifying and characterizing genes important in normal development and function of the ocular motility system, cranial nerves and brainstem and associated with congenital cranial dysinnervation disorders and related anomalies. | Ongoing
  This is an observational, descriptive study with no interventions geared towards identifying novel genes and characterizing their function, expression and impact on human cranial nerve development and disease. As genes previously undescribed in the human population are identified and characterized, reports regarding these details will be written and published but such timelines are impossible to predict. Also, as new information on previously identified genes is gathered generated, additional reports will be issued through scientific publications. As long as funding is available, the work will proceed in a rolling, ongoing timeline.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Engle, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JG, Tischfield MA, Nugent AA, Cheng L, Di Gioia SA, Chan WM, Maconachie G, Bosley TM, Summers CG, Hunter DG, Robson CD, Gottlob I, Engle EC. Loss of MAFB Function in Humans and Mice Causes Duane Syndrome, Aberrant Extraocular Muscle Innervation, and Inner-Ear Defects. Am J Hum Genet. 2016 Jun 2;98(6):1220-1227. doi: 10.1016/j.ajhg.2016.03.023. Epub 2016 May 12. PMID 27181683
- [Background] Balasubramanian R, Chew S, MacKinnon SE, Kang PB, Andrews C, Chan WM, Engle EC. Expanding the phenotypic spectrum and variability of endocrine abnormalities associated with TUBB3 E410K syndrome. J Clin Endocrinol Metab. 2015 Mar;100(3):E473-7. doi: 10.1210/jc.2014-4107. Epub 2015 Jan 5. PMID 25559402
- [Background] MacKinnon S, Oystreck DT, Andrews C, Chan WM, Hunter DG, Engle EC. Diagnostic distinctions and genetic analysis of patients diagnosed with moebius syndrome. Ophthalmology. 2014 Jul;121(7):1461-8. doi: 10.1016/j.ophtha.2014.01.006. Epub 2014 Mar 6. PMID 24612975
- [Background] Shaaban S, Ramos-Platt L, Gilles FH, Chan WM, Andrews C, De Girolami U, Demer J, Engle EC. RYR1 mutations as a cause of ophthalmoplegia, facial weakness, and malignant hyperthermia. JAMA Ophthalmol. 2013 Dec;131(12):1532-40. doi: 10.1001/jamaophthalmol.2013.4392. PMID 24091937
- [Background] Graeber CP, Hunter DG, Engle EC. The genetic basis of incomitant strabismus: consolidation of the current knowledge of the genetic foundations of disease. Semin Ophthalmol. 2013 Sep-Nov;28(5-6):427-37. doi: 10.3109/08820538.2013.825288. PMID 24138051
- [Background] Tischfield MA, Baris HN, Wu C, Rudolph G, Van Maldergem L, He W, Chan WM, Andrews C, Demer JL, Robertson RL, Mackey DA, Ruddle JB, Bird TD, Gottlob I, Pieh C, Traboulsi EI, Pomeroy SL, Hunter DG, Soul JS, Newlin A, Sabol LJ, Doherty EJ, de Uzcategui CE, de Uzcategui N, Collins ML, Sener EC, Wabbels B, Hellebrand H, Meitinger T, de Berardinis T, Magli A, Schiavi C, Pastore-Trossello M, Koc F, Wong AM, Levin AV, Geraghty MT, Descartes M, Flaherty M, Jamieson RV, Moller HU, Meuthen I, Callen DF, Kerwin J, Lindsay S, Meindl A, Gupta ML Jr, Pellman D, Engle EC. Human TUBB3 mutations perturb microtubule dynamics, kinesin interactions, and axon guidance. Cell. 2010 Jan 8;140(1):74-87. doi: 10.1016/j.cell.2009.12.011. PMID 20074521
- [Background] Miyake N, Andrews C, Fan W, He W, Chan WM, Engle EC. CHN1 mutations are not a common cause of sporadic Duane's retraction syndrome. Am J Med Genet A. 2010 Jan;152A(1):215-7. doi: 10.1002/ajmg.a.33168. No abstract available. PMID 20034095
- [Background] Di Gioia SA, Connors S, Matsunami N, Cannavino J, Rose MF, Gilette NM, Artoni P, de Macena Sobreira NL, Chan WM, Webb BD, Robson CD, Cheng L, Van Ryzin C, Ramirez-Martinez A, Mohassel P, Leppert M, Scholand MB, Grunseich C, Ferreira CR, Hartman T, Hayes IM, Morgan T, Markie DM, Fagiolini M, Swift A, Chines PS, Speck-Martins CE, Collins FS, Jabs EW, Bonnemann CG, Olson EN; Moebius Syndrome Research Consortium; Carey JC, Robertson SP, Manoli I, Engle EC. A defect in myoblast fusion underlies Carey-Fineman-Ziter syndrome. Nat Commun. 2017 Jul 6;8:16077. doi: 10.1038/ncomms16077. PMID 28681861
- [Background] Telegrafi A, Webb BD, Robbins SM, Speck-Martins CE, FitzPatrick D, Fleming L, Redett R, Dufke A, Houge G, van Harssel JJT, Verloes A, Robles A, Manoli I, Engle EC; Moebius Syndrome Research Consortium; Jabs EW, Valle D, Carey J, Hoover-Fong JE, Sobreira NLM. Identification of STAC3 variants in non-Native American families with overlapping features of Carey-Fineman-Ziter syndrome and Moebius syndrome. Am J Med Genet A. 2017 Oct;173(10):2763-2771. doi: 10.1002/ajmg.a.38375. Epub 2017 Aug 4. PMID 28777491
- [Background] Whitman MC, Miyake N, Nguyen EH, Bell JL, Matos Ruiz PM, Chan WM, Di Gioia SA, Mukherjee N, Barry BJ, Bosley TM, Khan AO, Engle EC. Decreased ACKR3 (CXCR7) function causes oculomotor synkinesis in mice and humans. Hum Mol Genet. 2019 Sep 15;28(18):3113-3125. doi: 10.1093/hmg/ddz137. PMID 31211835
- [Background] Grant PE, Im K, Ahtam B, Laurentys CT, Chan WM, Brainard M, Chew S, Drottar M, Robson CD, Drmic I, Engle EC. Altered White Matter Organization in the TUBB3 E410K Syndrome. Cereb Cortex. 2019 Jul 22;29(8):3561-3576. doi: 10.1093/cercor/bhy231. PMID 30272120
- [Background] Shaaban S, MacKinnon S, Andrews C, Staffieri SE, Maconachie GDE, Chan WM, Whitman MC, Morton SU, Yazar S, MacGregor S, Elder JE, Traboulsi EI, Gottlob I, Hewitt AW; Strabismus Genetics Research Consortium; Hunter DG, Mackey DA, Engle EC. Genome-Wide Association Study Identifies a Susceptibility Locus for Comitant Esotropia and Suggests a Parent-of-Origin Effect. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):4054-4064. doi: 10.1167/iovs.18-24082. PMID 30098192
- [Background] Di Gioia SA, Shaaban S, Tuysuz B, Elcioglu NH, Chan WM, Robson CD, Ecklund K, Gilette NM, Hamzaoglu A, Tayfun GA, Traboulsi EI, Engle EC. Recessive MYF5 Mutations Cause External Ophthalmoplegia, Rib, and Vertebral Anomalies. Am J Hum Genet. 2018 Jul 5;103(1):115-124. doi: 10.1016/j.ajhg.2018.05.003. Epub 2018 Jun 7. PMID 29887215
- [Background] Thomas MG, Maconachie GDE, Constantinescu CS, Chan WM, Barry B, Hisaund M, Sheth V, Kuht HJ, Dineen RA, Harieaswar S, Engle EC, Gottlob I. Congenital monocular elevation deficiency associated with a novel TUBB3 gene variant. Br J Ophthalmol. 2020 Apr;104(4):547-550. doi: 10.1136/bjophthalmol-2019-314293. Epub 2019 Jul 13. PMID 31302631
- [Background] Heidary G, Mackinnon S, Elliott A, Barry BJ, Engle EC, Hunter DG. Outcomes of strabismus surgery in genetically confirmed congenital fibrosis of the extraocular muscles. J AAPOS. 2019 Oct;23(5):253.e1-253.e6. doi: 10.1016/j.jaapos.2019.05.018. Epub 2019 Sep 18. PMID 31541710
- [Background] Sadeghi N, Hutchinson E, Van Ryzin C, FitzGibbon EJ, Butman JA, Webb BD, Facio F, Brooks BP, Collins FS, Jabs EW, Engle EC, Manoli I, Pierpaoli C; Moebius Syndrome Research Consortium. Brain phenotyping in Moebius syndrome and other congenital facial weakness disorders by diffusion MRI morphometry. Brain Commun. 2020;2(1):fcaa014. doi: 10.1093/braincomms/fcaa014. Epub 2020 Feb 14. PMID 32328577
- [Background] Webb BD, Manoli I, Engle EC, Jabs EW. A framework for the evaluation of patients with congenital facial weakness. Orphanet J Rare Dis. 2021 Apr 7;16(1):158. doi: 10.1186/s13023-021-01736-1. PMID 33827624
- [Background] Jurgens JA, Barry BJ, Lemire G, Chan WM, Whitman MC, Shaaban S, Robson CD, MacKinnon S, England EM, McMillan HJ, Kelly C, Pratt BM; Care4Rare Canada Consortium; O'Donnell-Luria A, MacArthur DG, Boycott KM, Hunter DG, Engle EC. Novel variants in TUBA1A cause congenital fibrosis of the extraocular muscles with or without malformations of cortical brain development. Eur J Hum Genet. 2021 May;29(5):816-826. doi: 10.1038/s41431-020-00804-7. Epub 2021 Mar 1. PMID 33649541